CLINICAL TRIAL: NCT01349777
Title: Effectiveness of Clopidogrel Resinate(PRegrel®) in Patients Undergoing Percutaneous Coronary Intervention Compared With ClopiDogrEl Bisulfate(Plavix®)
Brief Title: Effectiveness of Clopidogrel Resinate in PCI(PRIDE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-0483
Record Dates: First submitted 2011-04-22; First posted 2011-05-09 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease
Keywords: antiplatelet therapy post drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregrel® (Experimental): clopidogrel
  Interventions: Drug: Pregrel®
- Plavix® (Active Comparator): clopidogrel
  Interventions: Drug: Plavix®

INTERVENTIONS:
Drug: Pregrel® — Pregrel® 75mg daily for 12 months
  Other Names: clopidogrel
  Arms: Pregrel®
Drug: Plavix® — Plavix® 75mg daily for 12 months
  Other Names: clopidogrel 75mg
  Arms: Plavix®

SUMMARY:
This study is an open label, multi-center, randomized trial, which is designed to evaluate the efficacy and safety of clopidogrel derivative (Pregrel®) therapy for 12 months in patients undergoing PCI compared to conventional clopidogrel (Plavix®).

DETAILED DESCRIPTION:
Prospective, two arms, randomized multi-center trial of 1,056 patients enrolled at 3 centers in Korea.

Following angiography, patients with significant diameter stenosis >50% by visual estimation have documented myocardial ischemia or symptoms of angina and eligible for stenting without any exclusion criteria will be randomized 1:1 to: a) Pregrel® group vs. b) Plavix®. This trial is the non-inferiority study to demonstrate that the incidence of 12 months primary end-point in Pregrel® group.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Patients with symptomatic coronary artery disease with objective evidence of ischemia (e.g. symptoms of angina pectoris, positive stress test results, or dynamic ECG changes).
* Patients are referred for PCI, or thought to be at high likelihood for requiring stent placement with or without conventional balloon angioplasty
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:

  * Heparin
  * Aspirin
  * Both Clopidogrel and Ticlopidine
  * Stainless steel and/or
  * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenylhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled).
* Coronary anatomy not amenable to stent placement
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
* An elective major surgical procedure is planned that would necessitate interruption of thienopyridines during the first 1 year post enrollment.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Administration of the following medications prior to randomization: GpIIb-IIIa inhibitor and clopidogrel within 7 days (already received pretreatment), or thrombolytics within 24 hours.
* Long-term (at least > 3 months) use or requirement of NSAID or anticoagulation
* Patients with cardiogenic shock
* Acute MI patients within symptom onset < 12 hours needing primary angioplasty
* Patients with left main stem stenosis (>50% by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Actual)
Dates: Start 2010-03-15 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
composite of death (all cause-mortality), MI (Q wave and non Q wave) and stroke | 12 months

SECONDARY OUTCOMES:
composite of death, MI, stroke, or urgent revascularization | 12 months
Individual components of death, MI, stroke, or urgent revascularization | at discharge
The need for target vessel revascularization or any revascularization | 12 months
The incidence of early discontinuation of study drugs | 30 days
The incidence of major bleeding events | 30 days
Stent thrombosis | 30 days
composite of death, MI, stroke, or urgent revascularization | 30 days
composite of death, MI, stroke, or urgent revascularization | 6 months
Individual components of death, MI, stroke, or urgent revascularization | 30 days
Individual components of death, MI, stroke, or urgent revascularization | 6 months
Individual components of death, MI, stroke, or urgent revascularization | 12 months
The incidence of major bleeding events | 6 months
The incidence of major bleeding events | 12 months
The incidence of early discontinuation of study drugs | 6 months
The incidence of early discontinuation of study drugs | 12 months
Stent thrombosis | 6 months
Stent thrombosis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Gangneung Asan Hospital, Gangneung
  - Asan Medical Center, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.